CLINICAL TRIAL: NCT01202721
Title: Beta Blockers and Angiotensin Receptor Blockers in Bicuspid Aortic Valve Disease Aortopathy (BAV Study)
Acronym: BAV
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Terminated early due to lack of study feasibility and poor patient recruitment
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Population Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BAV-15JUNE2010
Record Dates: First submitted 2010-09-14; First posted 2010-09-16 (Estimated); Results first posted 2019-09-18 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-08

CONDITIONS: Cardiac Disease
Keywords: Congenital; Aortic Valve; Bicuspid; Aortopathy; bicuspid aortic valve aortopathy
MeSH Terms: conditions — Heart Diseases; Bicuspid Aortic Valve Disease | interventions — Atenolol; Telmisartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atenolol (Experimental): Atenolol or matching placebo 25 mg up-titrated to 100 mg.
  Interventions: Drug: Atenolol
- Telmisartan (Experimental): Telmisartan or matching placebo 40 mg up-titrated to 80mg
  Interventions: Drug: Telmisartan

INTERVENTIONS:
Drug: Atenolol — Atenolol or matching placebo 25 mg up-titrated to 100 mg
  Other Names: Atenolol 25/50/100 mg; or matched placebo
  Arms: Atenolol
Drug: Telmisartan — Telmisartan or matching placebo 40 mg up-titrated to 80mg.
  Other Names: Micardis 40/80 mg; or matched placebo
  Arms: Telmisartan

SUMMARY:
The purpose of this study is to determine whether long-term treatment with a beta-blocker (BB) such as atenolol and/or an angiotensin receptor blocker (ARB) such as telmisartan, given to adult patients with bicuspid aortic valve (BAV) disease (aortopathy) reduces the widening (dilatation) of the aorta from its baseline size.

DETAILED DESCRIPTION:
Bicuspid aortic valve (BAV) is the most common congenital heart disease lesion with an estimated 280 000 to 560 000 people affected in the Canada. Dilatation of the ascending aorta is a common feature in patients with BAV and is a result of inherent vascular abnormalities with superimposed effects of age and acquired cardiovascular risk factors. Severe aortic dilatation (> 50mm) leads to aortic dissection and premature death.

Histopathological studies of the aortas in patients with BAVs report similar findings to that of patients with Marfan syndrome. Beta Blocker (BB) therapy and more recently, Angiotensin Receptor Blocker (ARB) therapy, have been shown to decrease to rate of aortic dilatation and be of benefit to patients with Marfan syndrome. There is no such data however in patients with BAV and aortopathy.

Within the context of a randomized clinical trial, the investigators proposed to test the hypothesis that BB or ARB will reduce the rate of progressive aortic dilatation in adults with BAVs and ascending aortopathy as compared to placebo.

Design: Multicentre, randomized, double-blind, placebo-controlled, trial of adult patients with bicuspid aortic valve aortopathy. Patients who are eligible to take either study medication will be randomly allocated to participate in either the BB (atenolol) vs. placebo arm, or the ARB (telmisartan) vs. placebo arm. Patients who are ineligible for the BB arm will be assigned to the ARB vs. placebo arm and patients who are ineligible for the ARB arm will be assigned to the BB vs. placebo arm. Within each arm, all participants will be randomized to take either placebo or active medication. The atenolol arm will be up-titrated to100mg/day and the telmisartan arm will be up-titrated to 80 mg/day, or to the maximum tolerated dose.

ELIGIBILITY:
Inclusion Criteria:

* Age => 18 years
* Men and women with BAV and ascending aorta measuring > 37mm.
* Written informed consent

General Study Exclusion Criteria

1. History of cardiac diseases, such as

   * Symptomatic aortic stenosis or aortic regurgitation referred for surgical intervention or asymptomatic severe aortic stenosis or regurgitation based on current guidelines
   * Uncontrolled heart failure, right ventricular failure due to pulmonary hypertension
   * Cardiogenic shock
2. Systolic blood pressure < 100 mmHg
3. History of drug sensitivity, contraindication or adverse reaction to both BB and ARB. Participants who are able to tolerate only a BB will be allocated to the BB vs. placebo arm, and participants who are able to tolerate only an ARB will be allocated to the ARB vs. placebo arm, assuming no other exclusion criteria are met.
4. Ascending aorta measuring ≥ 50mm, requiring prophylactic ascending aorta surgery
5. Unable to provide informed consent
6. Need for both BB and ARB for treatment of concomitant medical conditions for which there are no other alternatives. Participants who are taking an ARB which cannot be discontinued will be allocated to the BB arm, and participants who are taking a BB which cannot be discontinued will be allocated to the ARB arm, if no other exclusion criteria are met.
7. Prior surgery on ascending aorta or aortic root (balloon valvuloplasty, aortic valvotomy or post coarctation surgery are acceptable)
8. Women who are pregnant at screening visit
9. Contraindication to MRI (claustrophobia, pacemaker, metallic clip in eye or brain)
10. History of any illness which limits the participants' ability to complete the study

Additional Exclusion Criteria for BB arm only

1. Heart rate <60 bpm
2. Heart block (1st, 2nd and 3rd degree AV block on ECG), or sick sinus syndrome
3. Asthma of sufficient severity to represent a contraindication to BB use in the judgment of the patient's physician
4. History of severe peripheral artery disorders
5. History of pheochromocytoma without the use of alpha-adrenergic blockers
6. History of metabolic acidosis

Additional Exclusion Criteria for ARB arm only

1. Women who are pregnant, lactating or who intend to become pregnant during the course of the study
2. Women who are of childbearing age and are not on reliable, accepted form of birth control
3. Hyperkalemia [serum potassium > 5.5 mmol/L] or renal dysfunction [GFR<45% measured by MDRD)
4. Patients being treated with an ACE Inhibitor that cannot be discontinued. (These patients may be randomized in the BB arm if no exclusion criteria are met.)
5. History of bilateral renal artery stenosis or unilateral renal artery stenosis to a solitary kidney
6. History of hepatic insufficiency and hepato-biliary obstruction
7. History of fructose intolerance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2016-04-19 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith Therrien, MD, Principal Investigator — MdGill University
Locations (13):
- Canada (13):
  - Mazankowski Alberta Heart Institute, Edmonton, Alberta
  - University of British Columbia, Vancouver, British Columbia
  - St. Boniface Hospital, Winnipeg, Manitoba
  - Hamilton Health Sciences-General, Hamilton, Ontario
  - Population Health Research Institute - Coordinating Centre, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Toronto General Hospital/University of Toronto, Toronto, Ontario
  - Cité de la Santé de Laval, Laval, Quebec
  - McGill University Health Centre, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec
  - Regina General Hospital, Regina, Saskatchewan

RESULTS

PARTICIPANT FLOW:
Groups:
- Atenolol: Atenolol 25 mg up-titrated to 100 mg.
- Telmisartan: Telmisartan 40 mg up-titrated to 80mg
- Atenolol Placebo: Participants in Atenolol group, randomized to receive matching placebo
- Telmisartan Placebo: Participants in Telmisartan group, randomized to receive matching placebo
Period: Overall Study
Arm/Group | Atenolol | Telmisartan | Atenolol Placebo | Telmisartan Placebo
Started | 18 | 26 | 14 | 27
Completed | 18 | 26 | 14 | 27
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Atenolol Placebo: Participants randomized to receive Atenolol placebo
- Telmisartan Placebo: Participants randomized to receive Telmisartan placebo
- Total: Total of all reporting groups
Arm/Group | Atenolol | Telmisartan | Atenolol Placebo | Telmisartan Placebo | Total
Number analyzed (Participants) | 18 | 26 | 14 | 27 | 85
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.4 (12.8) | 47 (12.2) | 49.1 (13.6) | 49.1 (11.2) | 47.3 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 8 | 7 | 27
  Male | 13 | 19 | 6 | 20 | 58
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  South Asian | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 1 | 1 | 0 | 4
  Black African | 0 | 0 | 0 | 1 | 1
  European | 15 | 23 | 12 | 26 | 76
  Native North American | 0 | 0 | 0 | 0 | 0
  Other | 1 | 2 | 1 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Ascending Aorta Size, as Evaluated by MRI
Description: The primary analyses include the evaluation of the effects of monotherapy (atenolol vs. placebo, telmisartan vs. placebo) on the change in aortic root size measured at 3 years. Change is measured in centimeters squared (final measurement - baseline measurement). Original outcome measure time frame was scheduled for 5 years, however due to poor study participant and site recruitment study was closed early and final outcome measures taken at approximately 3 years.
Time Frame: The difference between baseline measures (2012-2013) and Year 3 measure (2015-2016)
Population: Intention to treat analysis method followed: patients completed final visit over the phone where aortic root size cannot be measured; patients refused a final visit, or patient's information was received through a third party. Patients missing primary outcome measures still followed for other analyses.
Measure: Mean (Standard Deviation); unit: centimeters squared
Arm/Group | Atenolol | Telmisartan | Atenolol Placebo | Telmisartan Placebo
Number analyzed (Participants) | 16 | 23 | 13 | 25
centimeters squared | .6 (1.4) | .4 (1.3) | .7 (.8) | 1 (1.6)

2. Secondary Outcome: Rate of Change in Ascending Aorta Size Evaluated by Transthoracic Echocardiography (TEE)
Description: Rate of change in ascending aorta size evaluated by transthoracic echocardiography (ECHO) at 3 years. Change is measured in centimeters squared (final measurement - baseline measurement). Time frame was scheduled for 5 years, however due to poor study participant and site recruitment study was closed early and final outcome measures taken at approximately 3 years.
Time Frame: The difference between baseline measures (2012-2013) and Year 3 measure (2015-2016)
Population: Discrepancy exists between participant flow numbers and patients analyzed for the following reasons: patients completed final visit over the phone where aortic root size cannot be measured; patients refused a final visit, patient's information was received through a third party. Pt's not removed as they are still included in other analyses
Measure: Mean (Standard Deviation); unit: centimetres squared
Arm/Group | Atenolol | Telmisartan | Atenolol Placebo | Telmisartan Placebo
Number analyzed (Participants) | 17 | 21 | 12 | 23
centimetres squared | -.9 (3.2) | -.2 (4.5) | -1.6 (4.3) | .3 (2.8)

ADVERSE EVENTS:
Arm/Group | Atenolol | Telmisartan | Atenolol Placebo | Telmisartan Placebo
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/26 | 0/14 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/18 | 2/26 | 1/14 | 2/27
Other Adverse Events (participants affected / at risk) | 10/18 | 13/26 | 10/14 | 18/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Atenolol (N=18) | Telmisartan (N=26) | Atenolol Placebo (N=14) | Telmisartan Placebo (N=27)
Unexpected Serious Adverse Event (General disorders) | 0 | 2 | 1 | 2 — The adverse events were determined not unexpected and not related to study medication. They were related to serious but expected progression of disease or medical history. Specific organ system and adverse term event not specified in outcome analysis
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Atenolol (N=18) | Telmisartan (N=26) | Atenolol Placebo (N=14) | Telmisartan Placebo (N=27)
Chest Pain (Cardiac disorders) | 3 | 3 | 1 | 2
Shortness of Breath (Cardiac disorders) | 3 | 1 | 1 | 4
Dizziness (Vascular disorders) | 3 | 6 | 4 | 4
Syncope (Vascular disorders) | 0 | 0 | 0 | 1
Other (Investigations) | 1 | 3 | 4 | 7 — Other issues not listed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No